CLINICAL TRIAL: NCT07037914
Title: The Impact of the Nurse-Led "My Baby is Safe" Educational Program on Mothers' Knowledge, Skills, and Self-Efficacy
Brief Title: The Impact of the Nurse-Led "My Baby is Safe" Educational Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Dilara AYDIN TOZLU, Research Asssistant, Nurse, Amasya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13062025
Record Dates: First submitted 2025-06-13; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Sudden Infant Death Syndrome; Shaken Baby Syndrome
Keywords: Sudden Infant Death Syndrome; Shaken Baby Syndrome; Safe Sleep; Pediatric Nursing; Education
MeSH Terms: conditions — Sudden Infant Death; Shaken Baby Syndrome | interventions — Educational Status; Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Group I-Education and Counseling (Experimental)
  Interventions: Behavioral: Education and Counseling
- Control: Group II-Leaflet (Other)
  Interventions: Other: Leaflet

INTERVENTIONS:
Behavioral: Education and Counseling — The researcher will inform the mothers (n=25) that the My Baby is Safe Educational Program will be delivered individually through distance education via Microsoft Teams at times convenient for them, and that the program will be completed over 5 days. The scheduling will ensure that all modules included in the My Baby is Safe Educational Program are completed within one week at the latest. Mothers will be informed that they can receive telephone counseling from the researcher until their infants reach two months of age, and the researcher's phone number will be provided to them. During this period, the researchers will send weekly reminder messages to the mothers' phones, encouraging them to read the provided educational booklet and to watch the educational videos.
  The researcher will maintain communication with the mothers and conduct a home visit on the 15th day postpartum. During this home visit, the researcher will assess the infant's sleep environment for safe sleep practices.
  Arms: Experimental: Group I-Education and Counseling
Other: Leaflet — No structured or planned education will be provided to the control group by the researchers during the study period. After the first assessment, the mothers in the control group will receive a brochure prepared by the researchers based on the literature, containing brief informational notes on SIDS and SBS.
  The researcher will maintain communication with the mothers and conduct a home visit on the 15th day postpartum. During this visit, the researcher will observe the home environment where the infant resides and evaluate the infant's sleep environment in terms of safe sleep practices.
  After data collection from the intervention group has been completed, the same intervention (My Baby is Safe Educational Program) will also be delivered to the mothers in the control group.
  Arms: Control: Group II-Leaflet

SUMMARY:
The aim of this study is to determine the effect of the My Baby is Safe Educational Program on mothers' knowledge, skills, and self-efficacy levels.The objectives of the study are to ensure that mothers acquire sufficient knowledge and skills regarding SIDS and SBS, and to enhance their self-efficacy levels.The participants were randomly assigned to one group that received only the My Baby is Safe Educational Program (Group I), or to another group that received standard care (Group II).

DETAILED DESCRIPTION:
The aim of this randomized controlled study was to determine the effectiveness of the My Baby is Safe Educational Program on mothers' knowledge, skills, and self-efficacy related to the prevention of Sudden Infant Death Syndrome (SIDS) and Shaken Baby Syndrome (SBS).

This study, which included postpartum mothers, was conducted at Amasya University between July 2025 and July 2026. Participants were randomly assigned to either the intervention group, which received the My Baby is Safe Educational Program (Group I), or the control group, which received standard care (Group II).

The intervention consisted of a nurse-led, individualized, repetitive educational program that began in the postpartum period and included home visits. The program aimed to inform mothers about risk and protective factors for SIDS and SBS, to encourage the creation and maintenance of a safe sleep environment, and to promote the use of appropriate soothing techniques for crying infants.

The study sample consisted of 50 mothers, with 25 mothers assigned to each group. Data collection instruments included: the Infant and Parent Information Form, Sudden Infant Death Syndrome Awareness Scale - Mother Form, the Sudden Infant Death Syndrome Care Skills Form, the Shaken Baby Syndrome Awareness Assessment Scale-Short Form, the Shaken Baby Syndrome Care Skills Form, the Sleep Environment Checklist, and the Perceived Maternal Parenting Self-Efficacy Scale.

Data were analyzed using the licensed Statistical Package for the Social Sciences (SPSS v.23) software of Akdeniz University. Repeated measures ANOVA was used to evaluate the changes over time between the groups and the interaction effects between group and time. Spearman correlation analysis was performed to assess relationships between variables. The significance level was set at p<0.05. Additionally, effect sizes were calculated.

As a result, it is anticipated that the My Baby is Safe Educational Program will improve mothers' knowledge, skills, and self-efficacy related to the prevention of SIDS and SBS.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older,
* Having a healthy newborn,
* Having one or more children,
* Having at least a primary school education,
* Having a smartphone and mobile internet access,
* Being able to speak, read, listen, and understand Turkish, able to follow instructions, and having no communication barriers,
* Voluntarily agreeing to participate in the study.

Exclusion Criteria:

* Mothers whose newborns have any health problems will be excluded from the study.
* Mothers who wish to withdraw from the study at any point during the research process will be removed from the study.
* did not complete the process of the assessment and intervention of this study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Sudden Infant Death Syndrome Awareness | baseline (first assessment)
  Sudden Infant Death Syndrome Awareness Scale - Mother Form The scale consists of six items, divided into two sub-dimensions. These dimensions are 'Baby's Sleep Area' and 'Baby's Sleep Environment.' The scale uses a five-point Likert scale (Never = 1, Rarely = 2, Sometimes = 3, Often = 4, Always = 5). The last three questions of the scale are reverse-coded. The scale is interpreted based on the total scores of the subscales rather than the total score. As the score obtained from each subscale increases, it is interpreted that the level of awareness is also low. The Cronbach's alpha and McDonald's omega values for the 'Baby's Sleep Area' and 'Baby's Sleep Environment' subscales were found to be above 0.60.
Sudden Infant Death Syndrome Awareness | at the end of the invervention program (8 weeks after from baseline)
  Sudden Infant Death Syndrome Awareness Scale - Mother Form The scale consists of six items, divided into two sub-dimensions. These dimensions are 'Baby's Sleep Area' and 'Baby's Sleep Environment.' The scale uses a five-point Likert scale (Never = 1, Rarely = 2, Sometimes = 3, Often = 4, Always = 5). The last three questions of the scale are reverse-coded. The scale is interpreted based on the total scores of the subscales rather than the total score. As the score obtained from each subscale increases, it is interpreted that the level of awareness is also low. The Cronbach's alpha and McDonald's omega values for the 'Baby's Sleep Area' and 'Baby's Sleep Environment' subscales were found to be above 0.60.
Sudden Infant Death Syndrome Care Skills | baseline (first assessment)
  Sudden Infant Death Syndrome Care Skills Form (SIDS-CSF) The SIDS-CSF was developed by the researchers to assess mothers' care skills related to Sudden Infant Death Syndrome (SIDS). The researchers created the SIDS-CSF based on a review of the relevant literature. The form consists of a total of 28 items. It is structured as a 5-point Likert-type scale (Always, Frequently, Occasionally, Rarely, Never).
Sudden Infant Death Syndrome Care Skills | a home visit on the 15th day postpartum (2 weeks after from baseline)
  Sudden Infant Death Syndrome Care Skills Form (SIDS-CSF) The SIDS-CSF was developed by the researchers to assess mothers' care skills related to Sudden Infant Death Syndrome (SIDS). The researchers created the SIDS-CSF based on a review of the relevant literature. The form consists of a total of 28 items. It is structured as a 5-point Likert-type scale (Always, Frequently, Occasionally, Rarely, Never).
Sudden Infant Death Syndrome Care Skills | at the end of the invervention program (8 weeks after from baseline)
  Sudden Infant Death Syndrome Care Skills Form (SIDS-CSF) The SIDS-CSF was developed by the researchers to assess mothers' care skills related to Sudden Infant Death Syndrome (SIDS). The researchers created the SIDS-CSF based on a review of the relevant literature. The form consists of a total of 28 items. It is structured as a 5-point Likert-type scale (Always, Frequently, Occasionally, Rarely, Never).
Shaken Baby Syndrome Awareness | baseline (first assessment)
  Shaken Baby Syndrome Awareness Assessment Scale - Short Form (SBS-AAS-SF) The scale consists of three dimensions: soothing techniques, discipline techniques, and potential injury. The items in the scale are designed to assess whether the actions of caregivers are appropriate within each of these three dimensions. The scale includes 12 items for each dimension, totaling 36 items, and is formatted as a 6-point Likert scale. The correlations between the scores of the subscales indicate the degree of linearity among the three dimensions. The scale scores provide insight into the interrelationships of the constructs associated with shaking a baby, offering information on how effective interventions should be structured.
Shaken Baby Syndrome Awareness | at the end of the invervention program (8 weeks after from baseline)
  Shaken Baby Syndrome Awareness Assessment Scale - Short Form (SBS-AAS-SF) The scale consists of three dimensions: soothing techniques, discipline techniques, and potential injury. The items in the scale are designed to assess whether the actions of caregivers are appropriate within each of these three dimensions. The scale includes 12 items for each dimension, totaling 36 items, and is formatted as a 6-point Likert scale. The correlations between the scores of the subscales indicate the degree of linearity among the three dimensions. The scale scores provide insight into the interrelationships of the constructs associated with shaking a baby, offering information on how effective interventions should be structured.
Shaken Baby Syndrome Care Skills | baseline (first assessment)
  Shaken Baby Syndrome Care Skills Form The SBS-CSF was developed by the researchers to assess mothers' care skills related to Shaken Baby Syndrome (SBS). The researchers created the SBS-CSF based on a review of the relevant literature. The form consists of a total of 13 items. It is structured as a 5-point Likert-type scale (Always, Frequently, Occasionally, Rarely, Never).
Shaken Baby Syndrome Care Skills | a home visit on the 15th day postpartum (2 weeks after from baseline)
  Shaken Baby Syndrome Care Skills Form The SBS-CSF was developed by the researchers to assess mothers' care skills related to Shaken Baby Syndrome (SBS). The researchers created the SBS-CSF based on a review of the relevant literature. The form consists of a total of 13 items. It is structured as a 5-point Likert-type scale (Always, Frequently, Occasionally, Rarely, Never).
Shaken Baby Syndrome Care Skills | at the end of the invervention program (8 weeks after from baseline)
  Shaken Baby Syndrome Care Skills Form The SBS-CSF was developed by the researchers to assess mothers' care skills related to Shaken Baby Syndrome (SBS). The researchers created the SBS-CSF based on a review of the relevant literature. The form consists of a total of 13 items. It is structured as a 5-point Likert-type scale (Always, Frequently, Occasionally, Rarely, Never).
Self-Efficacy | baseline (first assessment)
  The Perceived Maternal Parenting Self-Efficacy Questionnaire The scale consists of 20 items and 4 subdimensions. It includes 18 positively worded items, rated on a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). The scale comprises three subfactors: "mother-infant interaction" (items 1, 2, 4, 5, 6, 7, 8, 13, 18), "caregiving procedures" (items 3, 14, 15, 16, 17), and "belief in the ability to foster positive infant behavior" (items 9, 10, 11, 12). Higher total scores indicate higher levels of maternal self-efficacy. A total score is obtained by summing the scores of all items.
Self-Efficacy | at the end of the invervention program (8 weeks after from baseline)
  The Perceived Maternal Parenting Self-Efficacy Questionnaire The scale consists of 20 items and 4 subdimensions. It includes 18 positively worded items, rated on a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). The scale comprises three subfactors: "mother-infant interaction" (items 1, 2, 4, 5, 6, 7, 8, 13, 18), "caregiving procedures" (items 3, 14, 15, 16, 17), and "belief in the ability to foster positive infant behavior" (items 9, 10, 11, 12). Higher total scores indicate higher levels of maternal self-efficacy. A total score is obtained by summing the scores of all items.

SECONDARY OUTCOMES:
Sleep Environment | a home visit on the 15th day postpartum (2 weeks after from baseline)
  Sleep Environment Checklist The Sleep Environment Checklist was developed by the researchers based on the relevant literature to assess mothers' care skills and compliance with safe sleep practices. The checklist consists of a total of 14 items.

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya University, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on reasonable request